CLINICAL TRIAL: NCT04402281
Title: Use of Algorithm for Safer and More Efficient Decision Making in the ED
Brief Title: Use of suPAR Algorithm for the ED Decision Making
Acronym: EDsuPAR
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Marja Mäkinen, PhD, Helsinki University Central Hospital
Other Study IDs: §33, HUS/141/2020 14.4.2020
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2021-06

CONDITIONS: Critical Illness
Keywords: ED; Critical illness; Decision making; POC test; suPAR
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- suPAR algoritm control: Control arm (Meilahti hospital): Samples are collected and suPAR measured but no algorithm is implemented.
  Interventions: Diagnostic Test: suPAR algoritm
- suPAR algoritm intervention: Intervention arm (Jorvi Hospital).
  According the algorithm when admitting a patient with suPAR below 3 ng/ml, physician should answer the following question
  "Are you sure it is the right decision to admit this patient? Please discuss this with a senior physician".
  If discharging a patient with suPAR above 6 ng/ml, physician should answer the following question
  "Are you sure it is the right decision to discharge this patient? Please discuss this with a senior physician".
  Interventions: Diagnostic Test: suPAR algoritm

INTERVENTIONS:
Diagnostic Test: suPAR algoritm — All medical patients attending to the ED and who will have blood drawn for routine examination will be part of the study. In patients with low suPAR (green group, suPAR below 3 ng/ml) and in patients with high suPAR (red group, suPAR > 6 ng/mL) the Intervention will be carried out

SUMMARY:
Will the use of a clinical decision algorithm in the ED improve discharge or admission decisions.

DETAILED DESCRIPTION:
Background Crowding and readmissions are common challenges in Emergency departments across Europe. The decision whether to admit or discharge the patient is challenging and is often based on clinical signs and symptoms e.g. blood pressure, pulse, respiratory rate, oxygen saturation and temperature. But some patients are unnecessarily admitted and may have been better off if sent home. Other patients may be discharged without - and one out of five patients are readmitted within a month raising the question whether the patient should have been admitted at first presentation in the ED. suPAR is a strong prognostic biomarker measured routinely in acute medical patients in some emergency department (ED) settings.suPAR is a broadly applicable biomarker of risk, and it has been developed an algorithm for simple interpretation of suPAR in clinical decisions for the study.

Objective To evaluate the use of a clinical decision algorithm in the ED with the aim of improving discharge or admission decisions.

ELIGIBILITY:
Inclusion Criteria:

* All patients above 18 years
* who are having blood taken for biochemical analysis when attending the ED

Exclusion Criteria:

* Acute medical patients that do not have blood drawn for routine biochemical testing.
* Pregnant
* Under 18 years old
* Terminally ill patients.

Ages: 18 Years to 104 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients during the study period who signed the consent
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Discharges | 30 days
  Number of discharges from the ED within 24 hours

SECONDARY OUTCOMES:
Admissions | 30 days
  Number of admissions to hospital
Length of stay | 30 days
  Length of stay during admission
Readmissions | 1,7 and 30 days
  Number of readmissions
Mortality | 30 days
  Number of Mortality

OTHER OUTCOMES:
Economical savings | 30 days
  Amount of money

CONTACTS AND LOCATIONS:
Overall Officials: Maaret Castrén, Docent, Principal Investigator — Professor
Locations (1):
- Department of Emergency Medicine and Services, Helsinki University Hospital and Helsinki University, Helsinki, Finland, Helsinki, Helsinki Usimaa, Finland

IPD SHARING:
Plan to Share IPD: No